CLINICAL TRIAL: NCT04647500
Title: Effects of Modulation of the Dopaminergic System Using Methylphenidate on Memory and Executive Processes in Individuals With 22q11.2 Deletion Syndrome
Brief Title: Effects of Methylphenidate on Brain and Cognition in 22q11 Deletion Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Stephan Eliez, Principal Investigator, University of Geneva, Switzerland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PB_201601472
Record Dates: First submitted 2020-11-03; First posted 2020-12-01 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: 22q11.2 Deletion Syndrome
MeSH Terms: conditions — DiGeorge Syndrome | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Depending on medication history and current psychostimulant medication, participants are included either in the consumer group (composed of participants with ongoing methylphenidate treatment) or in the naïve group (composed of participants naïve to the molecule)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 22q11DS naive (Other): 22q11DS participants naive to methylphenidate
  Interventions: Drug: Concerta
- 22q11DS consumer (Other): 22q11DS participants with a prolonged treatment of methylphenidate
  Interventions: Drug: Concerta

INTERVENTIONS:
Drug: Concerta — Evaluation of a treatment of Concerta over a period of 13 days.

SUMMARY:
Chromosome 22q11.2 deletion syndrome (22q11DS) is a neurogenetic condition associated with a high risk of psychiatric disorders, including schizophrenia spectrum disorders. This population is characterized by a specific neurocognitive profile and atypical brain development. Methylphenidate is a psychostimulant used in the treatment of attention deficit with/without hyperactivity (ADHD). Although ADHD is one of the most important co-morbidities in 22q11DS, affecting 35-45% of patients, to date only two studies have focused on quantifying the efficacy of this treatment in this population. The objective of this study is to quantify the improvement in cognitive performance as well as the differences in brain connectivity associated with the methylphenidate molecule in a population at risk of cognitive impairment and the development of schizophrenia.

DETAILED DESCRIPTION:
This study aimed to investigate the effects of methylphenidate (Concerta ®) in patients with 22q11DS. Outcome is evaluated based on changes in clinical and cognitive measures as well as brain connectivity (with magnetic resonance imaging and electroencephalography). Treatment benefits are evaluated in an intra-subject design, i.e. performance with/without treatment are compared for each patient. Depending on medication history and current psychostimulant medication, participants are included either in the consumer group (composed of participants with ongoing methylphenidate treatment) or in the naïve group (composed of participants naïve to the molecule). To the naive participants the investigators prescribe a 13-day treatment of Concerta ® at a weight-adjusted dose of 0.7 mg/kg). The treatment phase begins with a lower introductory dose for the first 5 days before moving on to the weight-adjusted dose. The effect of treatment on cognitive measures is assessed on day 6, with memory monitoring on days 7 and 13. The treatment effect evaluated using clinical measures and questionnaires was conducted at the end of the treatment phase to ensure multiple opportunities for observation by the participant and caregivers. For consumer participants, the procedure was similar. For visits with methylphenidate, participants will be asked to take their usual prescription. In order to best follow the procedure of the naïve group, for the visits without methylphenidate, the consumer participants were asked to interrupt their usual prescription for 13 days. Since many participants usually interrupt their treatment during vacations or sometimes on weekends, compliance is not a barrier. For methylphenidate-free visits, a 5-day break prior to assessment with cognitive measures will be requested from each participant. Again, in order to ensure several opportunities for observation for the participant and caregivers, assessments with clinical measures and questionnaires will be conducted at the end of the break, on day 13.

The research hypothesis of this study is that methylphenidate treatment has a beneficial effect on clinical and cognitive performance. Scores in the tests evaluating these areas are expected to be significantly better than when the tests were administered in the absence of the substance. A change in brain connectivity is also expected when the drug is taken, tending towards a "normalization" of brain connectivity. Finally, to find the link between changes in cognitive measures and changes in brain connectivity is investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed 22q11DS diagnosis.
* Minimum age of 8 years or maximum age of 25 years and 11 months.
* Attention difficulties pointed out by parents and/or the participant.
* Sufficient verbal expression and comprehension skills to understand and follow instructions based on initial interview.

Exclusion Criteria:

* Participants younger than 8 years and older that 25 years and 11 months.
* Previous adverse experience with MPH
* Cardio-vascular diseases including rhythm disorders, severe hypertension, cardiac insufficiency, obliterating cardiac and peripheral arterial disease, preexisting cerebrovascular affections, hemodynamically significant congenital heart defect, channelopathies.
* For the naïve group only: corrected QT (QTc) distance at baseline electrocardiogram above 460 milliseconds or elongation at control electrocardiogram (Day 6 of treatment) superior to 30 milliseconds with functional complaint.
* Psychiatric affections including anxiety attack, psychic tension or restlessness, manic episode, marked psychotic symptoms, schizophrenia, borderline personality disorder, clinical depression (present or past), suicidal episode, diagnosis or family history of Tourette syndrome, alcohol or drug abuse.
* Other somatic affections including hyperthyroid, glaucoma, pheochromocytoma.
* Concurrent treatment with monoamine oxidase inhibitors or interruption less than 14 days before beginning of treatment.
* Pregnancy or breastfeeding.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Conners' Continuous performance test, third edition (CPT-3) | CPT-3 pre-treatment
  Participants are instructed to press a button every time a letter appeared on the screen, except for the letter X where participants had to withhold their answer. Variables of interest are Detectability, Omission, Commission, Perseveration, Hit Reaction Time, Hit Reaction time Standard Deviation, Variability, Hit Reaction Time Block Change and Hit Reaction Time Inter- Stimulus Intervals Change.
Conners' Continuous performance test, third edition (CPT-3) | CPT-3 6 days of treatment
  Participants are instructed to press a button every time a letter appeared on the screen, except for the letter X where participants had to withhold their answer. Variables of interest are Detectability, Omission, Commission, Perseveration, Hit Reaction Time, Hit Reaction time Standard Deviation, Variability, Hit Reaction Time Block Change and Hit Reaction Time Inter- Stimulus Intervals Change.
Conners' Continuous performance test, third edition (CPT-3) | CPT-3 one month after the end of treatment
  Participants are instructed to press a button every time a letter appeared on the screen, except for the letter X where participants had to withhold their answer. Variables of interest are Detectability, Omission, Commission, Perseveration, Hit Reaction Time, Hit Reaction time Standard Deviation, Variability, Hit Reaction Time Block Change and Hit Reaction Time Inter- Stimulus Intervals Change.
Stroop task | Stroop inhibition ratio pre-treatment
  To measure the cost of cognitive inhibition in time, an inhibition ratio score is computed by dividing the raw score from the Stroop condition (participants have to name the color of the ink even though the word spells a different color) by the raw score in the color naming condition (participants are instructed to name rectangles of colors as fast as possible). This score reflects the cognitive cost of inhibiting the reading process. A ratio value close to 1 indicates a lesser cost of inhibition.
Stroop task | Stroop inhibition ratio 6 days of treatment
  To measure the cost of cognitive inhibition in time, an inhibition ratio score is computed by dividing the raw score from the Stroop condition (participants have to name the color of the ink even though the word spells a different color) by the raw score in the color naming condition (participants are instructed to name rectangles of colors as fast as possible). This score reflects the cognitive cost of inhibiting the reading process. A ratio value close to 1 indicates a lesser cost of inhibition.
Stroop task | Stroop inhibition ratio one month after the end of treatment
  To measure the cost of cognitive inhibition in time, an inhibition ratio score is computed by dividing the raw score from the Stroop condition (participants have to name the color of the ink even though the word spells a different color) by the raw score in the color naming condition (participants are instructed to name rectangles of colors as fast as possible). This score reflects the cognitive cost of inhibiting the reading process. A ratio value close to 1 indicates a lesser cost of inhibition.
Letter-number sequencing | Letter-number Sequencing pre-treatment
  A working memory subtest of the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Intelligence Scale for Children (WISC) in which the participant must sequence a random order of numbers and letters. Specifically, the participant must first say the numbers in ascending order and then the letters in alphabetical order. Longest sequence of letters and numbers correctly ordered
Letter-number sequencing | Letter-number Sequencing 6 days of treatment
  A working memory subtest of the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Intelligence Scale for Children (WISC) in which the participant must sequence a random order of numbers and letters. Specifically, the participant must first say the numbers in ascending order and then the letters in alphabetical order. Longest sequence of letters and numbers correctly ordered
Letter-number sequencing | Letter-number Sequencing one month after the end of treatment
  A working memory subtest of the Wechsler Adult Intelligence Scale (WAIS) and the Wechsler Intelligence Scale for Children (WISC) in which the participant must sequence a random order of numbers and letters. Specifically, the participant must first say the numbers in ascending order and then the letters in alphabetical order. Longest sequence of letters and numbers correctly ordered
Color Trails test (CTT) | CTT flexibility ratio pre-treatment
  To measure the cost of task switching, a flexibility ratio was calculated to account for processing speed by dividing the time to complete part B (drawing a line between number following chronological order while alternating between colors) by time to complete part A (drawing a line between number following chronological order). Value closer to 1 indicate better flexibility.
Color Trails test (CTT) | CTT flexibility ratio 6 days of treatment
  To measure the cost of task switching, a flexibility ratio was calculated to account for processing speed by dividing the time to complete part B (drawing a line between number following chronological order while alternating between colors) by time to complete part A (drawing a line between number following chronological order). Value closer to 1 indicate better flexibility.
Color Trails test (CTT) | CTT flexibility ratio one month after the end of treatment
  To measure the cost of task switching, a flexibility ratio was calculated to account for processing speed by dividing the time to complete part B (drawing a line between number following chronological order while alternating between colors) by time to complete part A (drawing a line between number following chronological order). Value closer to 1 indicate better flexibility.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | CANTAB pre-treatment
  The Motor Screening test (MOT) is a training procedure designed screen for difficulties with vision, movement, or comprehension and ascertains that the subject can follow simple instructions, as well as familiarising them with the touch screen.
  Intra-Extra Dimensional Set Shift (IED) is a test of rule acquisition and reversal. It features visual discrimination and attentional set formation maintenance, shifting and flexibility of attention.
  Spatial Working Memory (SWM) is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. It is a self-ordered task, which also assesses heuristic strategy.
  Stop Signal Task (SST) is a classic stop signal response inhibition test, which uses staircase functions to generate an estimate of stop signal reaction time. This test gives a measure of an individual's ability to inhibit a prepotent response.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | CANTAB 6 days of treatment
  The Motor Screening test (MOT) is a training procedure designed screen for difficulties with vision, movement, or comprehension and ascertains that the subject can follow simple instructions, as well as familiarising them with the touch screen.
  Intra-Extra Dimensional Set Shift (IED) is a test of rule acquisition and reversal. It features visual discrimination and attentional set formation maintenance, shifting and flexibility of attention.
  Spatial Working Memory (SWM) is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. It is a self-ordered task, which also assesses heuristic strategy.
  Stop Signal Task (SST) is a classic stop signal response inhibition test, which uses staircase functions to generate an estimate of stop signal reaction time. This test gives a measure of an individual's ability to inhibit a prepotent response.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | CANTAB one month after the end of treatment
  The Motor Screening test (MOT) is a training procedure designed screen for difficulties with vision, movement, or comprehension and ascertains that the subject can follow simple instructions, as well as familiarising them with the touch screen.
  Intra-Extra Dimensional Set Shift (IED) is a test of rule acquisition and reversal. It features visual discrimination and attentional set formation maintenance, shifting and flexibility of attention.
  Spatial Working Memory (SWM) is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. It is a self-ordered task, which also assesses heuristic strategy.
  Stop Signal Task (SST) is a classic stop signal response inhibition test, which uses staircase functions to generate an estimate of stop signal reaction time. This test gives a measure of an individual's ability to inhibit a prepotent response.
15 signes & 15 words | 15 signes & 15 words pre-treatment
  15 signs & 15 words is a homemade episodic memory task inspired by the Rey Auditory Verbal Learning Test (Rey, 1958). Participants are required to learn 15 common French words and 15 signs (drawings made out of 1 or 2 basic geometrical forms). After delays of thirty minutes, one day, one week and one month, participants are asked to freely recall the words and the signs they remembered. They are also asked to recognize the target items form a list of distractors. Variables of interest are (1) learning score = Maximum number of items correctly recalled during learning divided by the number of trials to reach learning criterion. Low score indicates poor learning. (2) Retention % thirty minutes/on day/one week = Number of items recalled after each delay in time divided by the maximum of items recalled during learning. Low score indicates poor memory.
15 signes & 15 words | 15 signes & 15 words 6 days of treatment
  15 signs & 15 words is a homemade episodic memory task inspired by the Rey Auditory Verbal Learning Test (Rey, 1958). Participants are required to learn 15 common French words and 15 signs (drawings made out of 1 or 2 basic geometrical forms). After delays of thirty minutes, one day, one week and one month, participants are asked to freely recall the words and the signs they remembered. They are also asked to recognize the target items form a list of distractors. Variables of interest are (1) learning score = Maximum number of items correctly recalled during learning divided by the number of trials to reach learning criterion. Low score indicates poor learning. (2) Retention % thirty minutes/on day/one week = Number of items recalled after each delay in time divided by the maximum of items recalled during learning. Low score indicates poor memory.
15 signes & 15 words | 15 signes & 15 words one month after the end of treatment
  15 signs & 15 words is a homemade episodic memory task inspired by the Rey Auditory Verbal Learning Test (Rey, 1958). Participants are required to learn 15 common French words and 15 signs (drawings made out of 1 or 2 basic geometrical forms). After delays of thirty minutes, one day, one week and one month, participants are asked to freely recall the words and the signs they remembered. They are also asked to recognize the target items form a list of distractors. Variables of interest are (1) learning score = Maximum number of items correctly recalled during learning divided by the number of trials to reach learning criterion. Low score indicates poor learning. (2) Retention % thirty minutes/on day/one week = Number of items recalled after each delay in time divided by the maximum of items recalled during learning. Low score indicates poor memory.
ADHD symptoms | ADHD symptoms pre-treatment
  Diagnostic and Statistical Manual of Mental Disorders - fifth edition (DSM-V)
ADHD symptoms | ADHD symptoms 13 days of treatment
  Diagnostic and Statistical Manual of Mental Disorders - fifth edition (DSM-V)
ADHD symptoms | ADHD symptoms one month after the end of treatment
  Diagnostic and Statistical Manual of Mental Disorders - fifth edition (DSM-V)

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) T1-weighted | MRI T1-weighted pre-treatment
  T1 structural images are collected to obtain accurate measurements of regional developmental changes in cortical morphometry comprising estimates of cortical volume, thickness and surface area. An MPRAGE T1-weighted sequence is employed with the following parameters: TR = 2500 ms, TE = 3 ms, flip angle = 8°, matrix acquisition = 256 × 256, field of view = 23.5 cm, slice thickness = 3.2 mm, 192 slices.
Magnetic Resonance Imaging (MRI) T1-weighted | MRI T1-weighted 6 days of treatment
  T1 structural images are collected to obtain accurate measurements of regional developmental changes in cortical morphometry comprising estimates of cortical volume, thickness and surface area. An MPRAGE T1-weighted sequence is employed with the following parameters: TR = 2500 ms, TE = 3 ms, flip angle = 8°, matrix acquisition = 256 × 256, field of view = 23.5 cm, slice thickness = 3.2 mm, 192 slices.
Magnetic Resonance Imaging (MRI) T1-weighted | MRI T1-weighted one month after the end of treatment
  T1 structural images are collected to obtain accurate measurements of regional developmental changes in cortical morphometry comprising estimates of cortical volume, thickness and surface area. An MPRAGE T1-weighted sequence is employed with the following parameters: TR = 2500 ms, TE = 3 ms, flip angle = 8°, matrix acquisition = 256 × 256, field of view = 23.5 cm, slice thickness = 3.2 mm, 192 slices.
MRI Spectroscopy | MRI Spectroscopy pre-treatment
  Acquisition of Single-voxel MRI Spectroscopy investigates changes in excitatory/inhibitory balance throughout development. More in detail, a Works-In-Progress (WIP) SVS (Single Voxel Spectroscopy) spin-echo sequence is used provided by Siemens and designed for detecting the GABA (Gamma-AminoButyric Acid) 1H MRS signal at 3 ppm in brain. 3 ROIs are selected: Anterior cingulate cortex (voxel size: 15 x 35 x 40, 98 avg), right hippocampus (voxel size: 20 x 30 x 40, 150 avg) and temporal cortex (voxel size: 30 x 30 x 30, 120 avg) that are manually placed during each session. Each sequence lasts around 7 minutes and patients are allowed to watch a video of their choice during the acquisition.
MRI Spectroscopy | MRI Spectroscopy 6 days of treatment
  Acquisition of Single-voxel MRI Spectroscopy investigates changes in excitatory/inhibitory balance throughout development. More in detail, a Works-In-Progress (WIP) SVS (Single Voxel Spectroscopy) spin-echo sequence is used provided by Siemens and designed for detecting the GABA (Gamma-AminoButyric Acid) 1H MRS signal at 3 ppm in brain. 3 ROIs are selected: Anterior cingulate cortex (voxel size: 15 x 35 x 40, 98 avg), right hippocampus (voxel size: 20 x 30 x 40, 150 avg) and temporal cortex (voxel size: 30 x 30 x 30, 120 avg) that are manually placed during each session. Each sequence lasts around 7 minutes and patients are allowed to watch a video of their choice during the acquisition.
MRI Spectroscopy | MRI Spectroscopy one month after the end of treatment
  Acquisition of Single-voxel MRI Spectroscopy investigates changes in excitatory/inhibitory balance throughout development. More in detail, a Works-In-Progress (WIP) SVS (Single Voxel Spectroscopy) spin-echo sequence is used provided by Siemens and designed for detecting the GABA (Gamma-AminoButyric Acid) 1H MRS signal at 3 ppm in brain. 3 ROIs are selected: Anterior cingulate cortex (voxel size: 15 x 35 x 40, 98 avg), right hippocampus (voxel size: 20 x 30 x 40, 150 avg) and temporal cortex (voxel size: 30 x 30 x 30, 120 avg) that are manually placed during each session. Each sequence lasts around 7 minutes and patients are allowed to watch a video of their choice during the acquisition.
MRI Resting State | MRI resting state pre-treatment
  Functional MRI sequence without stimulation (resting-state fMRI) scans are employed to assess the longitudinal changes in regional activity and functional connectivity measured by BOLD signal fluctuations. During this sequence, the participants are asked to fix a white cross on a black background for 8 minutes and leave their thoughts wander. Simultaneous recording of physiological parameters (heart rate and respiration) are employed to account for possible artifacts. (Parameters: 200 blood-oxygenation-level-dependent (BOLD) images with TR = 2400 ms, TE = 30 ms, 38 axial slices, slice thickness = 3.2 mm, flip angle = 85°, acquisition matrix = 94 × 128, field of view = 96 × 128).
MRI Resting State | MRI resting state 6 days of treatment
  Functional MRI sequence without stimulation (resting-state fMRI) scans are employed to assess the longitudinal changes in regional activity and functional connectivity measured by BOLD signal fluctuations. During this sequence, the participants are asked to fix a white cross on a black background for 8 minutes and leave their thoughts wander. Simultaneous recording of physiological parameters (heart rate and respiration) are employed to account for possible artifacts. (Parameters: 200 blood-oxygenation-level-dependent (BOLD) images with TR = 2400 ms, TE = 30 ms, 38 axial slices, slice thickness = 3.2 mm, flip angle = 85°, acquisition matrix = 94 × 128, field of view = 96 × 128).
MRI Resting State | MRI resting state one month after the end of treatment
  Functional MRI sequence without stimulation (resting-state fMRI) scans are employed to assess the longitudinal changes in regional activity and functional connectivity measured by BOLD signal fluctuations. During this sequence, the participants are asked to fix a white cross on a black background for 8 minutes and leave their thoughts wander. Simultaneous recording of physiological parameters (heart rate and respiration) are employed to account for possible artifacts. (Parameters: 200 blood-oxygenation-level-dependent (BOLD) images with TR = 2400 ms, TE = 30 ms, 38 axial slices, slice thickness = 3.2 mm, flip angle = 85°, acquisition matrix = 94 × 128, field of view = 96 × 128).
MRI Diffusion weighted images | MRI DSI pre-treatment
  Diffusion weighted images (DWI) are acquired to examine the longitudinal changes in white matter integrity and to quantify changes in tracts connecting a priori defined regions of interest. The patient would be warned about a slightly louder sequence sound and will be asked to watch their preferred video or closes their eyes and relax during this last sequence.
  DSI parameters are number of directions = 137, b = 3000 s/mm2, TR = 5100 ms, TE = 80 ms, Voxel size= 1.6x1.6x1.6, field of view = 23.9 cm, 64 axial slices, slice thickness = 1.6 mm.
MRI Diffusion weighted images | MRI DSI 6 days of treatment
  Diffusion weighted images (DWI) are acquired to examine the longitudinal changes in white matter integrity and to quantify changes in tracts connecting a priori defined regions of interest. The patient would be warned about a slightly louder sequence sound and will be asked to watch their preferred video or closes their eyes and relax during this last sequence.
  DSI parameters are number of directions = 137, b = 3000 s/mm2, TR = 5100 ms, TE = 80 ms, Voxel size= 1.6x1.6x1.6, field of view = 23.9 cm, 64 axial slices, slice thickness = 1.6 mm.
MRI Diffusion weighted images | MRI DSI one month after the end of treatment
  Diffusion weighted images (DWI) are acquired to examine the longitudinal changes in white matter integrity and to quantify changes in tracts connecting a priori defined regions of interest. The patient would be warned about a slightly louder sequence sound and will be asked to watch their preferred video or closes their eyes and relax during this last sequence.
  DSI parameters are number of directions = 137, b = 3000 s/mm2, TR = 5100 ms, TE = 80 ms, Voxel size= 1.6x1.6x1.6, field of view = 23.9 cm, 64 axial slices, slice thickness = 1.6 mm.
Electroencephalography (EEG) resting state | EEG resting state pre-treatment
  All the EEG data are continuously recorded with a sampling rate of 1000 Hz using a 256-electrode Hydrocel cap referenced to the vertex (Cz). Resting-state data with closed eyes is acquired for 6 minutes.
Electroencephalography (EEG) resting state | EEG resting state 6 days of treatment
  All the EEG data are continuously recorded with a sampling rate of 1000 Hz using a 256-electrode Hydrocel cap referenced to the vertex (Cz). Resting-state data with closed eyes is acquired for 6 minutes.
Electroencephalography (EEG) resting state | EEG resting state one month after the end of treatment
  All the EEG data are continuously recorded with a sampling rate of 1000 Hz using a 256-electrode Hydrocel cap referenced to the vertex (Cz). Resting-state data with closed eyes is acquired for 6 minutes.
EEG auditory | EEG Auditory pre-treatment
  Auditory steady state response paradigm: sequences of 2 types of auditory stimuli are presented binaurally: a 100 ripple tones (40 Hz) and 10 semi-randomly intermixed flat tones (1000 Hz). Ripple tones are presented at about 93 dB and the flat tones at about 83 dB. Participants are asked to detect the flat tone, while the ripple tones entrained the neural gamma oscillatory response. The duration of the task is around 7 minutes.
EEG auditory | EEG Auditory 6 days of treatment
  Auditory steady state response paradigm: sequences of 2 types of auditory stimuli are presented binaurally: a 100 ripple tones (40 Hz) and 10 semi-randomly intermixed flat tones (1000 Hz). Ripple tones are presented at about 93 dB and the flat tones at about 83 dB. Participants are asked to detect the flat tone, while the ripple tones entrained the neural gamma oscillatory response. The duration of the task is around 7 minutes.
EEG auditory | EEG Auditory one month after the end of treatment
  Auditory steady state response paradigm: sequences of 2 types of auditory stimuli are presented binaurally: a 100 ripple tones (40 Hz) and 10 semi-randomly intermixed flat tones (1000 Hz). Ripple tones are presented at about 93 dB and the flat tones at about 83 dB. Participants are asked to detect the flat tone, while the ripple tones entrained the neural gamma oscillatory response. The duration of the task is around 7 minutes.
EEG visual | EEG Visual pre-treatment
  Visual inward moving grating task paradigm: participants are presented with 3 blocks of 80 trials, with each trial consisting of a circular sinewave grating that contracted toward central fixation. The task of the participants is to detect and respond by button press to a velocity increase of the stimulus, randomly occurring between 750 and 3000 ms. Feedback on performance is provided on every trial, shortly after the response onset terminated stimulus presentation. The duration of the task is around 21 minutes in 3 blocks.
EEG visual | EEG Visual 6 days of treatment
  Visual inward moving grating task paradigm: participants are presented with 3 blocks of 80 trials, with each trial consisting of a circular sinewave grating that contracted toward central fixation. The task of the participants is to detect and respond by button press to a velocity increase of the stimulus, randomly occurring between 750 and 3000 ms. Feedback on performance is provided on every trial, shortly after the response onset terminated stimulus presentation. The duration of the task is around 21 minutes in 3 blocks.
EEG visual | EEG Visual one month after the end of treatment
  Visual inward moving grating task paradigm: participants are presented with 3 blocks of 80 trials, with each trial consisting of a circular sinewave grating that contracted toward central fixation. The task of the participants is to detect and respond by button press to a velocity increase of the stimulus, randomly occurring between 750 and 3000 ms. Feedback on performance is provided on every trial, shortly after the response onset terminated stimulus presentation. The duration of the task is around 21 minutes in 3 blocks.
Behavior Rating Inventory of Executive Function (BRIEF) questionnaire | BRIEF pre-treatment
  Children and Adults version. This questionnaire provides an ecological assessment of EF, with a Global Executive Composite (GEC) score derived from the Behavioral Regulation Index (BRI) and Metacognitive Index (MI). The BRI includes subscales of Inhibition, Shifting, Emotional regulation and only in the adult-form, Self- monitoring. The MI includes subscales of Initiation, Working memory, Planning, Organization and Monitoring. Observations are reported using standardized scores (T-scores)
Behavior Rating Inventory of Executive Function (BRIEF) questionnaire | BRIEF 13 days of treatment
  Children and Adults version. This questionnaire provides an ecological assessment of EF, with a Global Executive Composite (GEC) score derived from the Behavioral Regulation Index (BRI) and Metacognitive Index (MI). The BRI includes subscales of Inhibition, Shifting, Emotional regulation and only in the adult-form, Self- monitoring. The MI includes subscales of Initiation, Working memory, Planning, Organization and Monitoring. Observations are reported using standardized scores (T-scores)
Behavior Rating Inventory of Executive Function (BRIEF) questionnaire | BRIEF one month after the end of treatment
  Children and Adults version. This questionnaire provides an ecological assessment of EF, with a Global Executive Composite (GEC) score derived from the Behavioral Regulation Index (BRI) and Metacognitive Index (MI). The BRI includes subscales of Inhibition, Shifting, Emotional regulation and only in the adult-form, Self- monitoring. The MI includes subscales of Initiation, Working memory, Planning, Organization and Monitoring. Observations are reported using standardized scores (T-scores)

OTHER OUTCOMES:
Sensory-motor conflict 1 | Synchrony condition pre-treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 1 | Synchrony condition 6 days of treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 1 | Synchrony condition one month after the end of treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 2 | Asynchrony condition pre-treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 2 | Asynchrony condition 6 days of treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.
Sensory-motor conflict 2 | Asynchrony condition one month after the end of treatment
  The task uses a robotic device altering sensorimotor processing in participants and inducing mild to moderate hallucinations (presence hallucinations - PH) and passivity experiences. Participants move with their hand a robotic device placed in front of them. A second robot placed behind them reproduced their movements, thus delivering tactile feedback on their back either synchronously (0ms between the movement and the touch, sync) or asynchronously (delay of 500ms, async). Participants rate the strength of robot-induced PH, passivity experiences that they felt during robot manipulation, and control items. Occurrence and severity of clinical symptoms are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Eliez, Professor, Principal Investigator — University of Geneva, faculty of medicine
Locations (1):
- Developmental imaging and psychopathology lab, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No